CLINICAL TRIAL: NCT03137979
Title: The Safety and Efficacy Evaluation of Gingiva Mesenchymal Stem Cells Transplantation in Chronic Periodontitis Patients
Brief Title: Gingiva Mesenchymal Stem Cells Treatment of Chronic Periodontitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of Cell Thearpy Center, the First Hospital of HebeiMU, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17277787D-PD
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Periodontitis
Keywords: Periodontitis; Gingiva mesenchymal stem cells
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: GMSCs and collagen scaffolds (Experimental): Patients in group A will receive GMSCs seeded into collagen scaffolds at the local periodontal defects immediately after open flap debridement.
  Interventions: Biological: GMSCs and collagen scaffolds
- Group B: collagen scaffolds (Experimental): Patients in group B will receive collagen scaffolds implantation at the local periodontal defects immediately after open flap debridement.
  Interventions: Biological: Collagen scaffolds
- Group C: comparator (Other): Patients in comparator group will only undergo an open flap debridement.
  Interventions: Procedure: Open flap debridement

INTERVENTIONS:
Biological: GMSCs and collagen scaffolds — Patients in this group were given GMSCs and collagen scaffolds.
  Arms: Group A: GMSCs and collagen scaffolds
Biological: Collagen scaffolds — Patients in this group were given collagen scaffolds.
  Arms: Group B: collagen scaffolds
Procedure: Open flap debridement — The patients in this group will only receive the treatment of open flap debridement.
  Arms: Group C: comparator

SUMMARY:
This study is to evaluate the safety and efficacy of Gingiva Mesenchymal Stem Cell Therapy for Chronic Adult Periodontitis.

DETAILED DESCRIPTION:
Periodontitis featured by the progressive destruction loss of support tissues around the teeth has become a prevalent disease affecting the life quality of the adults. Although conventional periodontal treatment including open flap debridement and drug support therapy display reduced pocket depth and inflammation, the functional regeneration of the lost tissue and the repair of alveolar bone are insufficient. Gingiva mesenchymal stem cells (GMSCs) are multipotent cells possess the capacity of multilineage differentiation and have become an attractive optional treatment method for the regeneration of periodontal tissues and function. Therefore, GMSCs will be selected as seed cells to treat periodontitis. This study will recruit 30 patients which will be divided into three groups. 10 patients in group A will receive GMSCs seeded into collagen scaffolds at the local periodontal defects immediately after open flap debridement. 10 patients in group B will only receive collagen scaffolds devoid of GMSCs after open flap debridement. 10 patients in group C will only undergo an open flap debridement. This study will test the safety and efficacy of GMSCs implantation in chronic adult periodontitis through alveolous bone reproduction and other clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with adult periodontitis .
2. The age is from 35 to 60 years old.
3. The bleeding and coagulation function is normal.
4. The liver function is normal.
5. Patients who are suitable for routine treatment of periodontal curettage and other early treatments.
6. Pathological lesion is stable after the routine treatments.
7. Patients with the probing depth ≥6 mm and attachment loss level≥ 3 mm.
8. X ray plates show no significant root furcation lesion appears in the diseased teeth and the infrabony pocket is not less than 4mm deep.
9. Patients with good oral hygiene and/or in whom the plaque control is maintained excellently under the instruction of oral hygiene.
10. Patients who show good compliance.
11. Patients with tooth mobility of degreeⅡor less and the width of attached gingiva is considered appropriate for the existing Guided Tissue Regeneration (GTR) .
12. Patients who have understand the purposes of this clinical trial and can make an independent decision to comply with trial requirements.

Exclusion Criteria:

1. Patients with disease of the kidney, liver, blood and/or circulatory system.
2. Patients with diabetes (the fasting plasma glucose level≥7.0mmol/l).
3. Patients who are receiving treatment of hypertension and/or epilepsy.
4. Patients with malignant tumour or the history of this.
5. Patients with the genetic background of the periodontitis.
6. Patients with bone metabolic diseases.
7. Patients in need of administration of adrenal cortical steroid within 4 weeks.
8. Patients with alcoholics.
9. Patients who smoke more than 10 pieces of cigarettes.
10. Patients who suffer from drug induced gingival hyperplasia.
11. Patients with acute symptom of periodontitis.
12. The bone destruction is larger than 2/3 of the root length or the mobility tooth is investigated of more than degree Ⅱ.
13. Patients who are either pregnant, possibly pregnant or breast-feeding, or who hope to become pregnant during the period of the trial.
14. Patients who are participating in in other research team of clinical trial.
15. Patients with mental or consciousness disorder.
16. Patients with a previous history of hypersensitivity to any biological active drugs.
17. Patients who have undergo periodontal treatment within six months.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The evaluation of alveolar bone regeneration | Baseline and Post cell transplantation: 1,3, 6months after intervention
  A increase in the height of alveolar bone in mm examined by computed tomography (CT)

SECONDARY OUTCOMES:
Probing pocket depth (PPD) | Baseline and Post cell transplantation: 3, 6 months after intervention.
  A reduced distance in mm between the gingival margin and the bottom was measured by a manual periodontal probe.
Attachment level (AL) | Baseline and Post cell transplantation: 3, 6 months after intervention.
  A reduced distance in mm from the bottom of the periodontal pocket to the dentinocemental junction was examined by a manual probe.
Gingival index (GI) | Baseline and Post cell transplantation: 3, 6 months after intervention.
  A decreased degree of GI measured by a manual periodontal probe which was divided into 4 grades: 0, 1, 2 and 3.
Tooth mobility degree (TMD) | Baseline and Post cell transplantation: 1,3, 6months after intervention
  A decrease of periotest value was measured by periotest to evaluate the tooth mobility changes.

OTHER OUTCOMES:
Adverse reaction | Post cell transplantation: 1, 3, 6 months
  Adverse reaction include temperature changes, allergy, nausea and so on 6 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Baoyong Yan, Doctor, Study Chair — Hebei Medical University; Guangshun Liu, Master, Study Director — The First Hospital of Hebei Medical University; Quanhai Li, Doctor, Study Director — The First Hospital of Hebei Medical University; Xianyun Wang, Doctor, Principal Investigator — The First Hospital of Hebei Medical University; Jinhong Zhang, Master, Principal Investigator — The First Hospital of Hebei Medical University; Yao Wang, Bachelor, Principal Investigator — the First Hospital of Hebei Medical UniversityT; Jun Zhang, Master, Principal Investigator — The First Hospital of Hebei Medical University; Xiangwei Ren, Master, Principal Investigator — The First Hospital of Hebei Medical University; Qianfeng Liu, Bachelor, Principal Investigator — The First Hospital of Hebei Medical University; Yongbin Di, Master, Principal Investigator — The First Hospital of Hebei Medical University; Boyu Liu, Bachelor, Principal Investigator — The First Hospital of Hebei Medical University; Fan Zhang, Bachelor, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No